CLINICAL TRIAL: NCT01208142
Title: Dynamic Splinting for Toe Walking: a Randomized, Controlled Study With Gait Analysis
Brief Title: Toe Walker Gait Trial
Acronym: TW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unrelated to trial
Sponsor: Dynasplint Systems, Inc. (Industry)
Collaborators: McMurry University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010.001
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Gait
Keywords: toe walker; Pediatric toe walking; ankle flexion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): 25 Control subjects will only receive SOC (a weekly standardized physical therapy and daily wear of an AFO).
  Interventions: Other: standard of care treatment
- Dynasplint (Experimental): 25 Patients will receive the standard of care as well as an Ankle Flexion Dynasplint
  Interventions: Device: Ankle Flexion Dynasplint

INTERVENTIONS:
Other: standard of care treatment — weekly standardized physical therapy and daily wear of an AFO
  Arms: Standard of care
Device: Ankle Flexion Dynasplint — Weekly standardized physical therapy, daily wear of an AFO and nightly wear of the ankle flexion Dynasplint
  Arms: Dynasplint

SUMMARY:
The purpose of this study is to examine the change in ankle plantar flexion while walking, following treatment with the Ankle Dorsiflexion Dynasplint (AFD) for children diagnosed as Toe Walkers.

For twelve weeks, patients will either receive the standard treatment or the same standard treatment and the Dynaslint worn at night.

ELIGIBILITY:
Inclusion Criteria:

* Toe Walking secondary to CP
* Idiopathic TW
* Inability to ambulate with initial heel-contact
* Inability to bear weight and stand flat-footed for over one minute
* Inability to stand or hop on one foot (symptomatic) for more than one minute

Exclusion Criteria:

* Acid Maltase Deficiency Myopathy
* Acute Paralytic Poliomyelitis
* Spinal Muscular Atrophy-all types
* Stroke, ischemic or hemorrhagic, all types
* Multiple Sclerosis
* Traumatic Brain Injury (including Shaken Baby Syndrome)
* Unilateral ROM deficits in Knee or Hip
* Previous Achilles Tendon lengthening surgery
* Hemiplegic Cerebral Palsy
* Muscular Dystrophy-all types

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in plantar flexion while ambulating | 12 weeks
  The primary endpoint or dependent variable of this study will be the change in excessive plantar flexion while ambulating. A repeated measures analysis of variance (ANOVA) will be performed to measure kinematic change in gait patterns calculated with an ambulation laboratory test.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - Texas Tech University Health Sciences Center, Lubbock, Texas

REFERENCES:
- [Background] Lundequam P, Willis FB. Dynamic splinting home therapy for toe walking: a case report. Cases J. 2009 Nov 10;2:188. doi: 10.1186/1757-1626-2-188. PMID 19946498
- [Background] Booth MY, Yates CC, Edgar TS, Bandy WD. Serial casting vs combined intervention with botulinum toxin A and serial casting in the treatment of spastic equinus in children. Pediatr Phys Ther. 2003 Winter;15(4):216-20. doi: 10.1097/01.PEP.0000096382.65499.E2. PMID 17057457
- [Background] Li S, Bishop M, Sensac C. The Effect of Botulinium Toxin Type A Combined with Physical therapy on Gait in Children with idiopathic Toe Walking. Pediatric Physical Therapy. 2004 16(1):59.
- [Background] Romkes J, Hell AK, Brunner R. Changes in muscle activity in children with hemiplegic cerebral palsy while walking with and without ankle-foot orthoses. Gait Posture. 2006 Dec;24(4):467-74. doi: 10.1016/j.gaitpost.2005.12.001. Epub 2006 Jan 18. PMID 16413188
- [Background] Brouwer B, Davidson LK, Olney SJ. Serial casting in idiopathic toe-walkers and children with spastic cerebral palsy. J Pediatr Orthop. 2000 Mar-Apr;20(2):221-5. PMID 10739286
- [Background] Mulligan H, Wilmshurst E. Physiotherapy assessment and treatment for an ambulant child with cerebral palsy after botox A to the lower limbs: a case report. Pediatr Phys Ther. 2006 Spring;18(1):39-48. doi: 10.1097/01.pep.0000202252.92562.4c. PMID 16508533
- [Background] Willis AW, Crowner B, Brunstrom JE, Kissel A, Racette BA. High dose botulinum toxin A for the treatment of lower extremity hypertonicity in children with cerebral palsy. Dev Med Child Neurol. 2007 Nov;49(11):818-22. doi: 10.1111/j.1469-8749.2007.00818.x. PMID 17979859
- [Background] Gage JR. The role of gait analysis in the treatment of cerebral palsy. J Pediatr Orthop. 1994 Nov-Dec;14(6):701-2. No abstract available. PMID 7814578
- [Background] Romkes J, Brunner R. Comparison of a dynamic and a hinged ankle-foot orthosis by gait analysis in patients with hemiplegic cerebral palsy. Gait Posture. 2002 Feb;15(1):18-24. doi: 10.1016/s0966-6362(01)00178-3. PMID 11809577
- [Background] Hicks R, Durinick N, Gage JR. Differentiation of idiopathic toe-walking and cerebral palsy. J Pediatr Orthop. 1988 Mar-Apr;8(2):160-3. PMID 3350949
- [Background] Galli M, Crivellini M, Santambrogio GC, Fazzi E, Motta F. Short-term effects of "botulinum toxin a" as treatment for children with cerebral palsy: kinematic and kinetic aspects at the ankle joint. Funct Neurol. 2001 Oct-Dec;16(4):317-23. PMID 11853322
- [Background] Ubhi T, Bhakta BB, Ives HL, Allgar V, Roussounis SH. Randomised double blind placebo controlled trial of the effect of botulinum toxin on walking in cerebral palsy. Arch Dis Child. 2000 Dec;83(6):481-7. doi: 10.1136/adc.83.6.481. PMID 11087280
- [Background] Hemo Y, Macdessi SJ, Pierce RA, Aiona MD, Sussman MD. Outcome of patients after Achilles tendon lengthening for treatment of idiopathic toe walking. J Pediatr Orthop. 2006 May-Jun;26(3):336-40. doi: 10.1097/01.bpo.0000217743.44609.44. PMID 16670545
- [Background] Weigl D, Copeliovitch L, Itzchak Y, Strauss S. Sonographic healing stages of Achilles tendon after tenomuscular lengthening in children with cerebral palsy. J Pediatr Orthop. 2001 Nov-Dec;21(6):778-83. PMID 11675554
- [Background] Gage JR. Gait analysis in cerebral palsy. London, Mac Keith Press; 1991
- [Background] Lai J, Jones M, Willis B. Efficacy of Dynasplint Splinting on PlantarflexionTone and Contracture Seen in CVA and TBI Subject: A Controlled Cross-Over Study. Arch Phys Med Rehabil. 2007 Oct;88(10)
- [Background] Willis B. Post-TBI Gait Rehabilitation. Applied Neurol. 2007 Jul;3(7):25-26.